CLINICAL TRIAL: NCT06469385
Title: Phase 1 First in Human Dose Escalation and Safety Study of Topical ENS-002 for Atopic Dermatitis in Adults
Brief Title: Topical ENS-002 for Atopic Dermatitis in Adults
Acronym: EnSync
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Planned safety, efficacy and proof of mechanism obtained
Sponsor: Concerto Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENS-002-01
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema
Keywords: Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema

STUDY DESIGN:
Intervention Model Description: 3 participants will be included in each of three cohorts of ENS-002.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ENS-002 (Experimental): ENS-002 lotion to be applied topically either once or twice per day depending on assigned study cohort.
  Cohort 1 - once daily dose (QD) of low dose ENS-002. This dose will be applied topically to a single target site once daily for 7 days.
  Cohort 2 - QD dose of high dose ENS-002 in subjects with mild, moderate or severe Atopic Dermatitis. This dose will be applied topically to all affected skin (excluding scalp, face, groin, genitalia) once daily for 14 days.
  Cohort 3 - twice daily (BID) dose of high dose ENS-002 in subjects with mild, moderate or severe Atopic Dermatitis applied topically to all affected skin (excluding scalp, face, groin, genitalia) twice daily for 14 days
  Interventions: Biological: ENS-002

INTERVENTIONS:
Biological: ENS-002 — Live biotherapeutic product (LBP) consisting of commensal, clonal, non-pathogenic bacteria.
  Low Dose ENS-002 High Dose ENS-002

SUMMARY:
The goal of this study is to determine the safety and effects of ENS-002, a live biotherapeutic product (LBP) consisting of commensal, clonal, non-pathogenic bacteria in participants with atopic dermatitis.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, study investigating ENS-002, a live biotherapeutic product (LBP) consisting of commensal, clonal non-pathogenic bacteria

The purpose of this dose escalation study is to determine the recommended Phase 2 dose (RP2D) of ENS-002 in participants with mild, moderate or severe atopic dermatitis.

Participation in this study will continue until dose limiting toxicity or therapy intolerance, or participant withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign an informed consent form (ICF).
2. Age 18 years or older on the day of signing the ICF.
3. Diagnosis of AD according to Hanifin and Rajka
4. Atopic dermatitis has been diagnosed and present for ≥ 6 months prior to the first planned ENS-002 administration.
5. EASI (Eczema Area and Severity Index) score of 5 to 7 (mild) or 7.1 to 21 (moderate), or ≥ 21.1 or severe at screening.
6. Mild, moderate or severe AD as scored by the IGA at screening and baseline For Cohort 1, in which only a single antecubital fossa or other body site lesion will be administered ENS-002, a target lesion IGA will be performed.
7. Body surface area involvement must be ≥ 2% for mild AD and >10% for moderate to severe AD (excluding scalp, face, groin, and genitalia) at both screening and baseline as estimated based on the rule of nines and/or the palmar rule. Participants who have only one or a limited number of areas affected by AD (eg, neck, antecubital fossa, hands/feet, or popliteal involvement), as long as these sites have at least moderate severity, may also be eligible even if they do not meet the minimum BSA required - these participants will need to be approved by the Concerto Medical Monitor.
8. Presence of specific bacteria via qPCR. Two affected skin sites will be sampled as part of the screening tests; if at least one of the affected skin sites contains the specified bacteria, the participant is eligible pending eligibility in all the other inclusion/exclusion criteria. If the qPCR test does not detect the specified bacteria, the participant is not eligible, but the bacteria skin swabs may be repeated. No more than 2 attempts to detect the specified bacterial colonization over 28 days may be made.
9. Acceptable screening laboratory values that are within normal limits or are not clinically significantly abnormal. If clinical significance is unclear, the investigator must consult with Concerto's medical monitor.

   * Complete blood count with WBC differential (including absolute values).
   * Chemistry panel including hepatic transaminases.
   * CRP.
   * Urinalysis.
   * 12-lead electrocardiogram.
   * For women of childbearing potential (WOCBP), serum and/or urine test consistent with a non-pregnant state.
10. If using an oral and/or topical H1 antihistamine for pruritus and/or insomnia, must have been on a stable dose and frequency for at least 14 days prior to screening and must continue at the same dose and frequency throughout the study.
11. Willing and able to complete once-daily electronic diary entries for the duration of the study.

Exclusion Criteria:

1. Has only facial AD.
2. Has more than 20 Geographic Body Site Areas (GBSA) if to be enrolled into Cohort 2 or more than 10 GBSA if to be enrolled in Cohort 3 that are affected by AD. These GBSA restrictions exclude face, scalp, genitalia, and groin lesions. If the total number of allowable GBSAs is exceeded, the participant may be allowed to enroll after discussion with the Concerto Medical Monitor, but these additional sites must not have ENS-002 applied.
3. Presence of non-AD dermatologic disorder(s) including, but not limited to, the following dermatitides: photodermatitis, allergic contact, infestations (including scabies), eczematous eruption (eg, secondary to calcium channel blockers), nummular, stasis, dermatitis herpetiformis, xerotic, widespread seborrheic, bullous pemphigoid (prodromal phase), eczematous psoriasis, or mycosis fungoides (Sezary syndrome).
4. Presence of idiopathic chronic eczematous eruption of aging - defined as new-onset, atopic-like dermatitis presenting in people > 50 years old with no history of childhood AD.
5. Presence of indwelling arterial or venous catheters.
6. Cardiac valve disease history or artificial valve or pacemaker in place.
7. Implanted devices/prostheses including, but not limited to, eye lens, knee, hip, dental implants (but not caps or crowns), etc. replacements.
8. History of Grade 2 or higher neutropenia or leukopenia (except for known benign neutropenia typical for Fy(a-b-) status [formerly known as benign ethnic neutropenia or BEN]).
9. Unwilling to stop hair removal by any method (including shaving, waxing, or depilatory creams) in ENS-002 administration body sites for 7 days prior to the first ENS-002 administration and for at least 7 days after the last ENS-002 administration.
10. Any significant breaks or cracks in the skin in the target areas of ENS-002 administration, including severe excoriations or open or weeping wounds suggestive of an active infection/increased susceptibility to infection.
11. Clinically significant immunodeficiency (congenital or acquired [including a history of treated or untreated HIV, malnutrition, chronic viral infection]).
12. Netherton syndrome or other genodermatoses resulting in a defective epidermal barrier.
13. Active malignancy or history of malignancy in the past 3 years (Exceptions: superficial skin cancers - squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ of the skin, curatively treated with cryosurgery or surgical excision only and indolent prostate cancer).
14. Clinically significant cardiovascular, liver, pulmonary, neurologic, metabolic, or kidney disease or any other comorbid medical, surgical, social, or psychiatric condition, that, in the opinion of the investigator, puts the participant at increased risk, might lead to study noncompliance, and/or confounds interpretation of safety and efficacy data.
15. Required to take immunosuppressive drugs (eg, including but not limited to chemotherapy, systemic corticosteroids [≥ 10 mg prednisone equivalent/day; allowed corticosteroids: inhaled, intra-articular, topical low- to mid-potency creams (and lotions, gels, foams, etc.); use of allowed topical corticosteroids only after discussion and agreement with Medical Monitor, or if systemic, permitted at doses intended only for adrenal replacement, or if ≥ 5 days prior to first ENS-002 administration, on a one-time basis as a prophylaxis for imaging procedures], anti-tumor necrosis factor, colchicine, hydroxychloroquine, sulfasalazine, dapsone, methotrexate, mycophenylate mofetil, azathioprine, anti-interluekin-6 (anti-IL-6) antibody, anti-IL-1 antibody, or anti-CD20 antibody).
16. Lives with or has frequent contact with individual(s) with implantable medical devices including, but not limited to, artificial eye lens, artificial joint, cardiac stents, indwelling venous or arterial catheters, cardiac valvular disease, or artificial valve in place; or who have severe skin barrier defects or known immunodeficiency (congenital or acquired [eg, treated or untreated HIV, malnutrition, chronic viral infections]). If there is any question on this exclusion criterion contact the Concerto medical monitor.
17. Received oral or systemic antibiotics within 21 days prior to screening.
18. Inability to tolerate > 7 days without topical AD treatments and topical antibiotics (prescription or over-the-counter [OTC]) or has had topical antibiotics ≤ 7 days prior to screening.

    Exceptions:

    allowed emollients and low- and mid-potency corticosteroid creams. Low- and mid-potency corticosteroid creams may be allowed without a washout, but only after discussion and agreement with Concerto Medical Monitor. Allowed emollients may be substituted for disallowed emollients during screening as long as this occurs at least 7 days before the planned first ENS-002 administration.
19. Therapy prior to the first planned dose of ENS-002 with one or more of the following:

    1. Systemic corticosteroids within 28 days
    2. Topical high-potency corticosteroids within 28 days
    3. Low- and mid-potency corticosteroid creams within 14 days. These may be allowed if the participant is on a stable dose and after discussion and agreement with the Concerto Medical Monitor.
    4. Topical phosphodiesterase inhibitors within 7 days
    5. Emollients within 7 days, other than those emollients allowed in this study. If a participant has used a product with a 7-, 14-, or 28-day eligibility limit, a minimum of a 7-, 14-, or 28-day washout, respectively, is required before the first planned dose of ENS-002.
20. Treatment with systemic therapies with anti-pruritic (eg, tricyclic antidepressants, sedatives, tranquilizers, marijuana or other cannabinoids, opioid receptor agonists/antagonists) or pruritus- inducing (eg, opioids, angiotensin-converting enzyme inhibitors, cocaine, antimalarials) potential within 28 days prior to the first planned dose of ENS-002.
21. Therapy within 28 days prior to the first planned dose of ENS-002 with any immuno-modulating agents (eg, cyclosporine, azathioprine, methotrexate), phototherapy, or indoor tanning.
22. Therapy within 56 days or 5 half-lives (whichever is longer) prior to the first planned dose of ENS-002 with investigational drugs or any Janus kinase inhibitors (JAKs).
23. Concurrent therapy with dupilumab, tralokinumab, or lebrikizumab is allowed as long as participant has been on a stable dose for

    ≥ 16 weeks prior to the first planned dose of ENS-002. If a participant was taking any of these agents but has stopped, then a 56-day or five half-lives (whichever is longer) period is required before the first planned dose of ENS-002.
24. Bleach baths within 30 days prior to the first planned dose of ENS-002.
25. Use of any live topical bacterial product (OTC products within 4 weeks or investigational bacteria within 365 days) prior to the first planned dose of ENS-002.
26. Allergic to any of the excipients in ENS-002 (pea hydrolysate, potassium phosphate dibasic, sodium chloride, yeast extract, water for injection, glycerol, and methylcellulose).
27. Unable to use at least 2 of the 6 rescue antibiotics that cover all 3 bacteria in ENS-002.
28. Pregnant or planning to attempt to become pregnant during this study, breast feeding, breast pumping, or planning to breast feed.
29. Participant with a pregnant or breastfeeding partner or a partner planning to attempt to become pregnant during the study.
30. Unable to demonstrate proper ENS-002 application technique despite proficiency training.
31. Any prior exposure to ENS-002.
32. Is biologically a WOCBP; eg, has not had a hysterectomy, has not been in menopause for at least one year, and cannot or is unable or unwilling to use highly effective birth control measures during this study and for 90 days after the last administration of ENS-002.
33. If biologically male and fertile, cannot donate sperm and must adhere to highly effective birth control measures during this study and for 90 days after the last administration of ENS-002.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Safety of ENS-002 total doses | Up to 43 days
  Incidence of adverse events after applying different total doses of ENS-002 as measured by clinical laboratory tests, vital signs and physical examination at end of treatment compared to baseline
Safety of ENS-002 dose frequency | Up to 43 days
  Incidence of adverse events after applying different dose frequencies of ENS-002 as measured by clinical laboratory tests, vital signs and physical examination at end of treatment compared to baseline
Safety of ENS-002 different dose durations | Up to 43 days
  Incidence of adverse events after applying different dose durations of ENS-002 as measured by clinical laboratory tests, vital signs and physical examination at end of treatment compared to baseline
Tolerability of ENS-002 total doses | Up to 43 days
  Evaluate the tolerability of different total doses of ENS-002 administration as measured by clinical laboratory tests, vital signs and physical examination at end of treatment compared to baseline
Tolerability of ENS-002 different dose frequencies | Up to 43 days
  Evaluate the tolerability of different dose frequencies of ENS-002 administration as measured by clinical laboratory tests, vital signs and physical examination at end of treatment compared to baseline
Tolerability of ENS-002 different dose durations | Up to 43 days
  Evaluate the tolerability of different dose durations of ENS-002 administration as measured by clinical laboratory tests, vital signs and physical examination at end of treatment compared to baseline
Recommended Phase 2 Dose (RP2D) | Up to 43 days
  Evaluate the safety of applying different total doses, dose frequencies, and durations of ENS-002 administration to determine a tentative recommended Phase 2 dose (RP2D).

SECONDARY OUTCOMES:
Levels of specified bacterial colonization on affected skin | Up to 43 days
  Measure levels of specified bacterial colonization on affected skin by quantitative polymerase chain reaction (qPCR).
Levels of specified bacterial colonization on non-affected skin | Up to 43 days
  Measure levels of specified bacterial colonization on non-affected skin at end of treatment compared to baseline by quantitative polymerase chain reaction (qPCR).
ENS-002 skin colonization | Up to 43 days
  Measure extent of ENS-002 skin colonization at end of treatment compared to baseline quantitative by polymerase chain reaction (qPCR).
Peak Pruritus Numerical Rating Scale (PPNRS) pruritus | Up to 43 days
  Determine effects of ENS-002 on pruritus by absolute and mean changes in PPNRS at end of treatment compared to baseline
Peak Pruritus Numerical Rating Scale (PPNRS) affected skin | Up to 43 days
  Determine effects of ENS-002 on affected skin area by absolute and mean changes in PPNRS at end of treatment compared to baseline
Peak Pruritus Numerical Rating Scale (PPNRS) severity | Up to 43 days
  Determine effects of ENS-002 on severity by absolute and mean changes in PPNRS at end of treatment compared to baseline
Severity of Pruritus Scale (SPS) pruritus | Up to 43 days
  Determine effects of ENS-002 on pruritus by absolute and mean changes in SPS at end of treatment compared to baseline
Severity of Pruritus Scale (SPS) affected skin | Up to 43 days
  Determine effects of ENS-002 on affected skin area by absolute and mean changes in SPS at end of treatment compared to baseline
Severity of Pruritus Scale (SPS) severity | Up to 43 days
  Determine effects of ENS-002 on severity by absolute and mean changes in SPS at end of treatment compared to baseline
Eczema Area and Severity Index (EASI) affected skin | Up to 43 days
  Determine effects of ENS-002 on affected skin area by absolute change and percent of participants with a ≥ 50%, ≥ 75%, or ≥ 90% reduction in EASI at end of treatment compared to baseline
Eczema Area and Severity Index (EASI) severity | Up to 43 days
  Determine effects of ENS-002 on severity by absolute change and percent of participants with a ≥ 50%, ≥ 75%, or ≥ 90% reduction in EASI at end of treatment compared to baseline
Investigator Global Assessment (IGA) 0 to 1 | Up to 43 days
  Determine percent of participants with an Investigator Global Assessment (IGA) of 0 or 1 at end of treatment compared to baseline
Investigator Global Assessment (IGA) absolute decrease of at least 2 points | Up to 43 days
  Determine percent of participants with an absolute decrease of at least 2 points for moderate atopic dermatitis (AD) in Investigator Global Assessment (IGA) at end of treatment compared to baseline
Body Surface Area (BSA) absolute change | Up to 43 days
  Absolute change from baseline in percent BSA affected
Body Surface Area (BSA) mean change | Up to 43 days
  Mean change from baseline in percent BSA affected
Changes in corticosteroid use by participants | Up to 43 days
  Determine type, potency and frequency of corticosteroid use
Changes in corticosteroid use for flares | Up to 43 days
  Determine number of participants resorting to corticosteroids for flares.
ENS-002 Administration Compliance - percentage of planned administrations | Up to 14 days
  Assess compliance of actual ENS-002 administrations as a percentage of planned administrations determined by counting used and unused vials and asking participants
ENS-002 Administration Compliance recorded in ePRO diary | Up to 14 days
  Assess compliance of actual ENS-002 administrations by directed questions as recorded in an electronic participant reported outcome (ePRO) diary.

OTHER OUTCOMES:
Changes in White Blood Count (WBC) in peripheral blood | Up to 43 days
  Assess blood samples for changes in white blood cell (WBC) count after ENS-002 administration
Changes in WBC subsets in peripheral blood | Up to 43 days
  Assess blood samples for changes in WBC subsets (eg, neutrophils, lymphocytes) after ENS-002 administration
Changes in C-Reactive Protein (CRP) in peripheral blood | Up to 43 days
  Assess blood samples for changes in CRP after ENS-002 administration
Changes in immune cells in peripheral blood | Up to 43 days
  Assess blood samples for changes in immune cells after ENS-002 administration
Changes in cytokines in peripheral blood | Up to 43 days
  Assess blood samples for changes in cytokines after ENS-002 administration
Changes in immunoglobulin E (IgE) in peripheral blood | Up to 43 days
  Assess blood samples for changes in immunoglobulin E (IgE) after ENS-002 administration
Changes in chemokines in peripheral blood | Up to 43 days
  Assess blood samples for changes in chemokines after ENS-002 administration
Changes in skin inflammatory markers | Up to 43 days
  Skin tape strips will be taken to assess changes in immune markers including cytokines and chemokines after ENS-002 administration
Microbiome changes on affected skin not administered ENS-002. Microbiome changes on affected and non-affected skin. | Up to 43 days
  Skin swabs to evaluate microbiome changes on affected skin that was not administered ENS-002
Microbiome changes on affected skin administered ENS-002. Microbiome changes on affected and non-affected skin. | Up to 43 days
  Skin swabs to evaluate microbiome changes on affected skin that was administered ENS-002
Microbiome changes on non-affected skin Microbiome changes on affected and non-affected skin. | Up to 43 days
  Skin swabs to evaluate microbiome changes on non-affected skin
Participant preferences and feedback on feasibility and tolerability of ENS-002 administration. | Up to 43 days
  Collect Electronic participant reported outcomes (ePRO). The ePRO diary will include specific questions on skin color change, pruritus, rash, pain, tenderness, fever, chills, night sweats, and other side effects, along with ease of application, skin feel, interference with use of emollients or other topically applied agents, effect on usual hygiene practices, residual feel after dosing has stopped, and effect on activities of daily living (eg, sleep, exercise, wearing clothing).

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Cervantes, PhD, Study Chair — Concerto Biosciences
Locations (3):
- United States (3):
  - Encore Medical Research, Hollywood, Florida
  - Northeast Dermatology Associates, Beverly, Massachusetts
  - Derm Research, Austin, Texas